CLINICAL TRIAL: NCT00671645
Title: Preoperative Combined RadioChemo-MolecularTargetTherapy of the Locally Advanced Rectum Carcinoma (cT3NxM0) - a Phase II Pilot Study With Preoperative Application of Capecitabine, Bevacizumab and Radiotherapy (RTx)
Brief Title: Preoperative Combined RadioChemo-Molecular Target Therapy With Capecitabine, Bevacizumab, and Radiotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: reaching of step 1 (recruitment of 8 patients) per protocol -> risk assessment -> termination because of occurance of toxicity Grade 3 and 4
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG R04/TAKO 08
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Rectal Cancer
Keywords: pilot study; rectal; carcinoma; phase II; preoperative; RadioChemo; molecular; target; therapy; T3; ABCSG; TAKO; R04; 08
MeSH Terms: conditions — Rectal Neoplasms; Carcinoma; Erythema Multiforme | interventions — Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: capecitabine, bevacizumab

INTERVENTIONS:
Drug: capecitabine, bevacizumab — Capecitabine 825 mg/m2 bid (on each therapy day of first 4 Therapy weeks) Bevacizumab 5 mg/kg weight; day 1, 15, 29
  Other Names: Xeloda; Avastin

SUMMARY:
* feasibility and tolerance of preoperative therapy with Bevacizumab in combination with Capecitabine and radiotherapy for patients with locally advanced, locally operable rectal carcinoma
* collection of response rate (T- and M-downstaging, pathological complete remission)

DETAILED DESCRIPTION:
Combined RadioChemotherapy:

Therapy start: within 28 days after bioptical diagnosis

Radiotherapy: 5 x 5 days 1.8 Gy radiotherapy; cummulative dose 45 Gy

Chemotherapy: Capecitabin 825mg/m² bid, on each radiation day during the first 4 weeks RCTx

Molecular Targeted Therapy: Bevacizumab 5 mg/kg body weight; day 1, 15, 29 Operation due to TME adherence to a break of min. 42 to max. 56 days after the last application of bevacizumab

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 80
* bioptical confirmed adenocarcinoma of the rectum in T3NxM0 status. The tumor has to be basically surgically complete resectable (->R0).
* no former chemotherapy, radiotherapy of pelvis or abdomen and/or tumor resection of rectum carcinoma
* WHO performance status 0-2
* adequate bone marrow reserve (granulocytes >= 3.000/µl, absolute neutrophil >= 0 1,5 x 10 9/l thrombocytes: >= 100.000/µl, haemoglobin >= 10g/dl)
* adequate hepatic function (Bilirubin: <= 1.5 x ULN, GOT und GPT <= 2.5 x ULN)
* adequate renal function (creatinin: <= 1.25 mg/dl, creatinin-clearance: > 50 ml/min (Cockcroft and Gault formula)), proteinuria: dipstick < 2+. In case of dipstick > 2+ protein has to be measured in 24h urine and does not exceed more than 1g/24h)
* ability of intake of pills
* women of childbearing potential: exclusion of pregnancy (negative urin or serum pregnancy test)
* willingness of women of childbearing potential and accordingly of potent men to use approved contraceptives (e.g. birth-control pill, loop, condom) during and at least 3 month after conclusion of the study
* life expectancy of at least 3 month
* INR and aPTT < 1.5 ULN
* signed Informed Consent before recruitment

Exclusion Criteria:

* failure of one inclusion criteria
* former radiotherapy of pelvis or abdomen
* former chemotherapy
* any other kind of malign tumor in the last 5 years
* any other kind of tumour in the last 5 years with exception of basal cell carcinoma of skin and cervix carcinoma in situ
* general contraindication or known hypersensitivity against Bevacizumab and/or Capecitabine
* non malign disease, if there is a contraindication with radiotherapy, or chemotherapy with Bevacizumab and Capecitabine, or a resection of rectum: uncontrolled hypertension (systolic > 150 mmHG and/or diastolic >100 mmHG) or clinical significant (e.g. active) cardiovascular disease: CVA (cardiovascular accident)/ cerebral apoplexy (< 6 months before recruitment), myocardial infarct (< 6 months before recruitment), instable angina pectoris, CHF with NYHA status II or higher, or treated serious arrhythmia, hepatic disease, significant neurologic or psychiatric disorders
* florid, serious infections at the time of recruitment
* peripheral neuropathy (NCI CTC >= Grade 1)
* legally limited contractual capability or evidence of neurological or psychiatric disease, if it will constrict the patients compliance in the opinion of the investigator
* evidence of lacking cooperation of the patient
* major intervention within 28 days before recruitment, open wounds
* serious injuries, unhealed wounds or fractures
* patients with spinal compressions or metastases in central nervous system
* evidence of bleeding diathesis or coagulation dysfunction
* actual intake of anticoagulant or thrombolytic agents, Aspirin > 325 mg/d or within 10 days before study start)
* actual or recent (within 10 days before recruitment) therapeutic therapy with fully-dosed anticoagulants. A prophylactic treatment is permitted.
* previous thromboembolic or hemorrhagic events within the last 6 months before recruitment
* previous abdominal fistulas, GI perforation or intra-abdominal abscess within the last 6 months
* treatment with other study medication within 28 days before recruitment
* patients with malabsorption syndrome or difficulties swallowing
* pregnant or breast feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02-27 (Actual); Study Completion 2009-02-27 (Actual)

PRIMARY OUTCOMES:
feasibility and tolerance of preoperative therapy with Bevacizumab in combination with Capecitabine and radiotherapy for patients with locally advanced, locally operable rectal carcinoma | descriptive evaluation

SECONDARY OUTCOMES:
collection of response rate (T- and M-downstaging, pathological complete remission) | descriptive evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Oefner, MD, MSc, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group; Alexander de Vries, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group; Wolfgang Eisterer, MD, Principal Investigator — ABCSG, TAKO
Locations (10):
- Austria (10):
  - Hospital BHB St. Veit/Glan, Surgery, Saint Veit/Glan, Carinthia
  - Medical University Graz, Oncology, Graz, Styria
  - State Hospital Leoben, Surgery, Leoben, Styria
  - Medical University Innsbruck, Internal Medicine, Innsbruck, Tyrol
  - Hospital BHS Linz, Radiooncology, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen, Coop. Group, Wels, Upper Austria
  - State Hospital Feldkirch, Radiotherapy, Feldkirch, Vorarlberg
  - State Hospital Salzburg-Paracelsius Medical University - Oncology, Salzburg
  - Hospital BHB Vienna, Surgery, Vienna
  - Medical University Vienna, Radiotherapy, Vienna

REFERENCES:
- See also: Related Info — http://www.abcsg.at